CLINICAL TRIAL: NCT02981693
Title: 1-year Evaluation of iRoot SP as a Root Canal Sealer Compare to AH Plus Sealer: A Prospective Clinical Study
Brief Title: Evaluation of iRoot SP as Root Canal Sealer: A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui Chen (Other)
Responsible Party: Sponsor-Investigator, Hui Chen, Professor, The Dental Hospital of Zhejiang University School of Medicine
Organization: The Dental Hospital of Zhejiang University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZhejiangU
Record Dates: First submitted 2016-11-27; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: Irreversible Pulpitis; Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- iRoot SP sealer (Experimental): iRoot SP sealer was used as root canal sealer in root canal obturation.
  Interventions: Procedure: Root canal sealer
- AH Plus sealer (Active Comparator): AH Plus sealer was used as a gold standard to be compared with iRoot SP sealer in root canal obturation.
  Interventions: Procedure: Root canal sealer

INTERVENTIONS:
Procedure: Root canal sealer — Patients who required root canal therapy were enrolled and allotted into either iRoot SP arm or AH Plus arm randomly.For Test Arm: iRoot SP was used as a sealer. Obturation was performed with Gutta-percha cones and root canal sealer by continuous-wave condensation technique. For Control Arm: AH Plus was used as root canal sealer. The same steps were followed for obturation as in Test Arm.

SUMMARY:
The purpose of this study was to evaluate the clinical and radiological outcomes of iRoot SP as a root canal sealer in comparison with AH Plus sealer within 1-year follow up.Patients needing root canal treatment were enrolled and allotted into either iRoot SP group or AH Plus arm randomly. After root canal shaping and cleaning, the teeth were obturated according to their arms. Assessment of postoperative pain was done 1 week after root canal obturation using visual analog scale. After 1-year follow-up, clinical and radiographic evaluations were carried out. Statistical analysis at P < 0.05 was conducted to measure difference between the arms.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to:

1. have a mature tooth with closed apices;
2. have one single or multi-rooted tooth with irreversible pulpitis, pulp necrosis or apical periodontitis;
3. be prepared to appear for follow-up and
4. sign informed consent form.

Exclusion Criteria:

Subjects with:

1. moderate or severe marginal periodontitis;
2. internal or external root resorption in periapical radiograph;
3. active systemic disease;
4. physical or mental disability,
5. pregnant or lactating

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Radiographical assessments | 1 year after root canal therapy
  The periapical status was assessed in the radiographs.Teeth with complete restitution of the periodontal contours were judged as "healed". Teeth with a clearly decreased size of the periapical radiolucency were judged as "healing". Teeth with unchanged, increased, or new periapical radiolucency were judged as "failed".

SECONDARY OUTCOMES:
Clinical assessments | 1 year after root canal therapy
  The root filled tooth was considered clinically successful if there was absence of clinical sign or symptom such as spontaneous pain, sensitivity to percussion or palpation, abnormal mobility, signs of pathology like abscess or sinus tract.
Postoperative Pain Evaluation | 1 week after root canal therapy
  Pain was evaluated by using a visual analogue scale (VAS) made of a 10 cm line, where 0 = no pain and 10 = unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, Study Chair — Affiliated Hospital of Stomatology, College of Medicine, Zhejiang University